CLINICAL TRIAL: NCT02407769
Title: Effect of a Late Evening Supplementation With Branched Chain Amino Acids on the Nutritional Status in Patients on the Waiting List for Liver Transplantation
Brief Title: Late Evening Supplementation With Branched Chain Amino Acids in Liver Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Guanajuato (Other)
Collaborators: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Niko Alain Cruz Sancén, Dietitian, Universidad de Guanajuato
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GAS-1103-13/14-1
Record Dates: First submitted 2015-03-17; First posted 2015-04-03 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Liver Cirrhosis
Keywords: Liver transplantation; Liver cirrhosis; Branched chain amino acids; Late evening supplementation; Nutritional status
MeSH Terms: conditions — Liver Cirrhosis | interventions — Amino Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Branched chain amino acids (Experimental): The patients will drink a Enterex Hepatic bag (500 Kcal, 18.6g of proteins of which 8.63g are branched chain amino acids, 71.7g of carbohydrates and 15.4g of lipids) during the late evening (after 19:00 hours) daily by two months.
  Interventions: Dietary Supplement: Late evening supplementation with branched chain amino acids
- Late evening snack (Sham Comparator): The patients will eat a snack with similar nutrimental facts that food supplement (480 Kcal, 19g of proteins and they were based in casein and vegetable proteins; 17g of lipids and 63g of carbohydrates) during the late evening (after 19:00 hours) daily by two months.
  Interventions: Dietary Supplement: Late evening supplementation with branched chain amino acids

INTERVENTIONS:
Dietary Supplement: Late evening supplementation with branched chain amino acids — The patients will drink a Enterex Hepatic bag (500 Kcal, 18.6g of proteins of which 8.63g are branched chain amino acids, 71.7g of carbohydrates and 15.4g of lipids) during late evening (after 19:00 hours) in comparison with the late evening snack group which will eat a snack based in food with the next nutrimental facts (480 Kcal, 19g of proteins based in casein and vegetables sources, 17g of lipids and 63g of carbohydrates) during the same schedule that intervention group.
  Other Names: Enterex hepatic

SUMMARY:
Assess the impact in body composition and handgrip strength of the nocturne supplementation by a month with BCAA (Enterex hepatic in patients awaiting liver transplantation)

DETAILED DESCRIPTION:
Clinical trial study was make, data were obtained from people awaiting liver transplantation and with at least a criteria of protein/energy malnutrition (fase angle < 5.4°, subjective global assessment B or C and/or handgrip strength < 30 in men and < 20 in women). The investigators make them body composition assessment (weight, height, body mass index [BMI], mean arm circumference [MAC], muscle arm area [MAA], tricipital skinfold, Dual X ray absorptiometry [fat mass and fat free mass]) and handgrip strength at beginning and after 30 days of nocturne supplementation with BCAA and standardized diet (35-40 Kcal, 55% carbohydrates, 25% lipids and 20% proteins).

ELIGIBILITY:
Inclusion Criteria:

* Patients on waiting list for liver transplantation.
* Diagnosis of undernutrition.

Exclusion Criteria:

* Hepatorrenal syndrome.
* Hepatopulmonar syndrome
* Diabetes
* Overweight

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in Body Composition | Basal and 30 and 60 days after intervention.
  The body composition will be measured with air displacement pletismografy through Bodpod the results will be expressed in percentaje of fat mass and fat free mass.

SECONDARY OUTCOMES:
Change in Mid arm muscle area | Basal and 30 and 60 days after intervention.
  Estimation of muscle area of the no dominant arm using the formula [(MAMA - (π x PT))2 / 4 π ]
  - 10 in men and -6.5 in women, the result is expressed in cm2.
Change in Quality of life | Basal and 30 and 60 days after intervention.
  It will be measured by the questionnaire SF-36 that is a generic scale providing a health profile and is applicable for both, patients and general population; the results that the 36 questions divided in 8 dimensions. The patients answers will be transformed to a numeric scale: since 0 (worst) to 100 (better)
Change in Fase angle. | Basal and 30 and 60 days after intervention.
  vectorial sum of the resistance and reactance result in the impedance, and the angle that is formed is called the fase angle; this is obtain through a impedanciometre, the measure is expressed in grades.
Change in Handgrip strength. | Basal and 30 and 60 days after intervention.
  Handgrip strength of the no dominant hand will be measured by a hand dynamometer in kilograms/Force

CONTACTS AND LOCATIONS:
Overall Officials: Niko Alain Cruz Sancén, Principal Investigator — Universidad de Guanajuato
Locations (1):
- Instituto Nacional de ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico City, Mexico